CLINICAL TRIAL: NCT05461248
Title: An Exploratory Study on the Recovery of Intestinal Flora and Intestinal Function by Preventing Stoma Discharge Reinfusion After Sphincter Preservation for Middle and Low Rectal Cancer
Brief Title: Stoma Discharge Reinfusion After Sphincter Preservation for Middle and Low Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STARS-RC04
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The experimental group collected stoma exudates and used an enema bag to infuse them from the anus.
  The control group was not reinfused.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The stoma drainage fluid was reinfused once a week for 2 months after radical rectal surgery. For each reinfusion, eat liquid food the day before, collect 400-600mL of stoma discharge on the same day (if the stoma fluid is too small, it can be mixed with warm water), and use an enema bag to reinfuse from the patient's anus. Generally, the flow rate is controlled at about 100mL/min.
  Interventions: Procedure: stoma drainage reinfusion
- Conventional group (Sham Comparator): The conventional group received no additional intervention.
  Interventions: Procedure: Standard of Care - No Return of Stoma Drain

INTERVENTIONS:
Procedure: stoma drainage reinfusion — 1 month after radical rectal surgery, the stoma drainage fluid was reinfused once a week for 2 months. For each reinfusion, eat liquid food the day before, collect 400-600mL of stoma discharge on the same day (if the stoma fluid is too small, it can be mixed with warm water), and use an enema bag to reinfuse from the patient's anus. Generally, the flow rate is controlled at about 100mL/min.
  Arms: Experimental group
Procedure: Standard of Care - No Return of Stoma Drain — No Return of Stoma Drain
  Arms: Conventional group

SUMMARY:
To analyze the occurrence of defecation complications, rectal function, and quality of life indicators after sphincter-preserving surgery for middle and low rectal cancer, the stoma exudate was collected before the stoma was restored, and the defecation complications, rectal function and quality of life indicators were evaluated. The effect of anal reinfusion of stoma discharge on the recovery of intestinal function in patients.

DETAILED DESCRIPTION:
Previous studies have shown that the mucosa and villi of the left intestinal segment will atrophy after intestinal bypass, the absorption capacity will decrease, and the rhythmic contraction will disappear. Some studies have shown that irrigation through the anorectal cavity may help prevent and treat colorectal anastomotic fistulas and improve the postoperative life of patients. Based on this, it is hypothesized that the stimulation of stomal exudate anal reinfusion to the empty intestinal segment through the anus may help to promote the recovery of intestinal function and intestinal flora disturbance after stoma retraction.

In response to this hypothesis, in this study, we intend to carry out a prospective and observational study on patients with stoma resection, aiming to investigate whether the stimulation of stoma discharge and anal reinfusion of stoma drainage through the anus before resection has any effect on the anus. It is beneficial to the recovery of intestinal function, reducing the occurrence of complications and improving the imbalance of intestinal flora, providing high-level clinical evidence.

ELIGIBILITY:
Inclusion criteria

1. Age: 18~75 years old, male or female;
2. Pathological diagnosis of adenocarcinoma of the rectum on preoperative biopsy;
3. Clinical staging was T1-4aN0-2M0;
4. No distant multiple metastases;
5. ECOG rating 0-2;
6. Cardiac, pulmonary, hepatic and renal functions met the criteria for surgical tolerance
7. Clinical diagnosis of middle and low rectal cancer, the lower edge of the tumour is within 10cm from the anal verge, and it is proposed to perform radical rectal surgery and prophylactic ileostomy at stage I, and intestinal closure at stage II;
8. Patients and their families were able to understand and willing to participate in this clinical study and signed an informed consent form.

Exclusion criteria

1. Previous history of malignant colorectal tumour or recently diagnosed combination of other malignant tumours; 2、Patients with combined intestinal obstruction, intestinal perforation, intestinal haemorrhage, etc. requiring emergency surgery; 3. Neighbouring organs requiring combined organ removal; 4. ASA classification ≥ Grade IV and/or ECOG physical status score > 2; 5. Those who have serious liver and kidney dysfunction, cardiopulmonary dysfunction, coagulation dysfunction or combined serious basic diseases cannot tolerate the surgery; 6. Have a history of serious mental illness; 7. Pregnant or breastfeeding women; 8. Those who have a history of taking steroid drugs; 9. Patients with other clinical and laboratory conditions considered by the investigator to be inappropriate for participation in the trial; 10. One week before the operation, there are signs of infection, body temperature rises >37.5°C, blood WBC >10.0×109/L; 11. History of antibiotic use 1 week prior to surgery (excluding preoperative shock medication); 12. Preoperative neoadjuvant patients

Exit criteria

1. Accompanied by other non-oncological conditions that make it impossible for the patient to continue to receive this treatment plan;
2. After enrolment in the study, patients who required emergency surgery due to intestinal obstruction, perforation, or bleeding,et al. prior to stoma closure;
3. Patients with pathologically confirmed distant metastases after rectal surgery, including liver, pelvis, ovary, peritoneum, and distant lymph node metastases;
4. Intraoperative exploration for middle and low rectal cancer in anus-preserving surgery for those who need combined organ resection;
5. After enrolment in the study, patients requested to withdraw from the study cohort for various reasons, or were unable to complete the study programme and follow-up for various reasons;
6. Anastomotic fistula, severe anastomotic stenosis (inability to pass through enteroscopy or oesophageal finger and inability to dilate via oesophageal finger) after radical rectal surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of low anterior resection syndrome | six months after stoma closure surgery
  Incidence of low anterior resection syndrome six months after stoma closure surgery

SECONDARY OUTCOMES:
Bacteriological sequencing after stoma closure surgery | 1 month after stoma reversal
  Bacteriological sequencing 1 month after stoma closure surgery
Low Anterior Resection Syndrome (LARS) questionnaire | 1 month after stoma reversal
  Low Anterior Resection Syndrome, is a clinical condition that occurs in patients who have undergone anterior resection of the rectum, resulting in bowel dysfunction and experience at least one of the symptoms associated with LARS, leading to at least one negative consequence. The LARS scale classifies patients into three severity categories: no LARS (0-20), mild LARS (21-29), and major LARS (30-42). Higher scores mean a worse outcome.
Wexner incontinence score | 1 month after stoma reversal
  The Wexner Incontinence Score, also known as the Wexner Constipation Grading Scale, is a quantitative tool used to assess the severity of anal incontinence. This scoring system calculates scores by patients completing a daily defecation questionnaire to assess their anal control function. The Wexner incontinence score typically covers the following aspects: gas incontinence, liquid fecal incontinence, solid fecal incontinence, use of liners, lifestyle changes. Each evaluation item has a corresponding score range, usually from 0 to 4 points, where 0 points means it never happened and 4 points means it always happened. Add up the scores of all projects to obtain the total score. The total score ranges from 0 to 20, with 0 indicating completely normal and 20 indicating the most severe incontinence.
MSKCC Bowl Function Questionnaire | 1 month after stoma reversal
  The MSKCC Bowl Function Questionnaire is a tool used to evaluate the intestinal function of patients with rectal cancer after undergoing surgery, radiation therapy, chemotherapy, and other treatments. This questionnaire typically contains multiple items, each asking questions about different aspects of the patient's intestinal function. Except for the first item, all other items are rated on a Likert 5-point scale, namely "always", "often", "sometimes", "rarely", and "never", with scores of 1, 2, 3, 4, and 5, respectively. In the questionnaire, certain items are set as reverse scoring, meaning that the higher the score, the worse the function. The total score of the scale is obtained by adding the scores of all items. The higher the total score, the better the patient's intestinal function. Due to the inclusion of reverse scoring items in the questionnaire, special treatment is required for these items when calculating the total score to ensure its accuracy and reliability.
Glazer pelvic floor muscle surface electromyography | 1 month after stoma reversal
  Glazer pelvic floor muscle surface electromyography is a detection method used to evaluate the function of pelvic floor muscles. This method collects electromyographic signals of pelvic floor muscles through surface electrodes, and then evaluates the functional status of pelvic floor muscles. By analyzing the amplitude, frequency, variability, and other parameters of these electrical signals, the supportive function, sexual function, and sphincter function of pelvic floor muscles can be evaluated. The evaluation process typically includes five stages: pre resting stage, phase contraction stage, tonic contraction stage, endurance contraction stage, and post resting stage. The higher the score, the better the pelvic floor muscle function. At the same time, it is necessary to assess the performance of pelvic floor muscles in different functional aspects based on individual scores.
Quality of life (QOL) score | 1 month after stoma reversal
  QOL score is often used to assess the quality of life and health status of a cancer patient, and based on these health status scores, determine the treatment options that the patient can accept. The evaluation indicators mainly include 12 aspects, including appetite, mental state, sleep, fatigue, pain, family understanding and cooperation, colleagues' understanding and cooperation, personal understanding of cancer, attitude towards treatment, daily life, side effects of treatment, and facial expressions. 60 points is the maximum score, if it is less than 20 points, it belongs to extremely poor quality of life; 21-30 points belong to poor quality of life; a score of 31-40 indicates an average quality of life; a score of 41-50 indicates a relatively good quality of life; a score of 51-60 indicates a good quality of life.
Recovery of postoperative bowel function | 1 month after stoma reversal
  After reversal surgery, time to oral feeding, time to anal defecation after reduction surgery, and rate of intestinal obstruction (intestinal obstruction was defined as ,inability to tolerate food for more than 72 H or the need for re-fasting or gastrointestinal decompression) were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Prof., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, He L, Zhang L, Sun J, Wang Y, Wang M, Zhao Y, Sun X, Gong Y, Li Z, Guo Y, Wang Q. Effects of stoma discharge reinfusion on low anterior resection syndrome and the gut microbiota following sphincter-preserving surgery for middle and low rectal cancer: a randomized clinical trial. Updates Surg. 2025 Nov 13. doi: 10.1007/s13304-025-02454-0. Online ahead of print. PMID 41233674

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT05461248/Prot_SAP_000.pdf